CLINICAL TRIAL: NCT06188910
Title: Effectiveness of a Neurofeedback Intervention on Symptoms of Anxiety and Psychological Distress Associated With Smartphone Use in Young Adults
Brief Title: Neurofeedback and Nomophobia in Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Salamanca (Other)
Collaborators: Instituto de Investigación Biomédica de Salamanca (Other); Gerencia Regional de Salud de Castilla y Leon (Other)
Responsible Party: Principal Investigator, José Ignacio Recio Rodriguez, Principal investigator, University of Salamanca
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IBYE23_00001 - GRS2709/A1/2023
Record Dates: First submitted 2023-12-18; First posted 2024-01-03 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Anxiety; Biofeedback
MeSH Terms: conditions — Anxiety Disorders | interventions — Neurofeedback; Biofeedback, Psychology

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Neurofeedback (Experimental): 3 weekly 30-minute neurofeedback sessions per week for 12 weeks
  Interventions: Other: Neurofeedback
- Control (Active Comparator): Health education, a 25-minute session, on mobile phone addiction and promotion of healthy lifestyles
  Interventions: Other: Health education

INTERVENTIONS:
Other: Neurofeedback — Conducting neurofeedback sessions guided by a researcher
  Other Names: Biofeedback
  Arms: Neurofeedback
Other: Health education — Health education on mobile phone addiction
  Arms: Control

SUMMARY:
Introduction: Given the growing increase in addiction to social networks and smartphone use in young people and its implications for health, it is necessary to investigate effective interventions for the appropriate use of these technologies and coping with possible signs of addiction.

Objective: To evaluate the effect of an intervention based on neurofeedback techniques on anxiety and other disorders associated with problematic use of mobile phones and the internet in young adults.

Methodology: Randomised controlled clinical trial with two parallel groups: an intervention group (IG) and a control group (CG). The study population will be young adults aged 18-30 years. A sample size of 40 participants has been estimated, 20 in each group to detect a difference of 3.9 points or more on the DASS-21 anxiety questionnaire.

All participants will receive an educational workshop on the responsible use of new technologies and the promotion of healthy lifestyles. The IG, in addition to this educational workshop, will receive 25 neurofeedback sessions during 12 weeks, 2-3 sessions/week with the MUSE neurofeedback device.

A baseline and 3-month post-intervention assessment will be conducted for both groups to study change variables related to smartphone addiction (Smartphone Addiction Scale-Short Version (SAS-SV)), nomophobia (Nomophobia Questionnaire (NMP-Q)), depression, anxiety and stress (Depression, Anxiety and Stress Scale 21-item (DASS-21)) and sleep quality.

ELIGIBILITY:
Inclusion Criteria:

* Have one or more mobile devices such as smartphones.
* Have a compatible mobile device to install and use the Muse: EEG Meditation & Sleep application.
* Be fully functional.
* Willingness to voluntarily participate in the study and sign the informed consent form.

Exclusion Criteria:

* History of severe psychiatric disorders (such as schizoaffective disorders, bipolar disorder, major depressive episode with symptoms or other non-organic psychotic disorders) requiring psychiatric treatment in the 6 months prior to study entry.
* History of brain injury or other problems contraindicating the use of neurofeedback.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Anxiety | Baseline, 3-months
  Anxiety evaluated through Depression, Anxiety and Stress Scale 21-item (DASS-21). Minimum 0 - maximum 63

SECONDARY OUTCOMES:
Nomophobia | Baseline, 3-months
  Nomophobia evaluated through Nomophobia Questionnaire (NMP-Q). Minimum 20 - maximum 140
Sleep Quality | Baseline, 3-months
  Sleep quality evaluated through Atenas questionnaire. Minimum 0 - maximum 24

CONTACTS AND LOCATIONS:
Overall Officials: José Ignacio Recio Rodriguez, PhD, Principal Investigator — University of Salamanca
Locations (1):
- University of Salamanca, Salamanca, Salamanca, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fernandez-Crespo M, Rihuete-Galve MI, Sanchez-Aguadero N, Sanchez-Sanchez N, Gonzalez-Sanchez J, Garcia-Yu IA, Lee HC, Recio-Rodriguez JI. Efficacy of neurofeedback-assisted mindfulness for anxiety and nomophobia in Spanish young adults: a randomized controlled trial. Front Public Health. 2025 Dec 2;13:1712564. doi: 10.3389/fpubh.2025.1712564. eCollection 2025. PMID 41409706
- [Derived] Fernandez-Crespo M, Recio-Rodriguez JI, Lee HC, Alonso-Dominguez R, Montejo AL, Hernandez-Gonzalez L, Iglesias Sierra V, Rihuete-Galve MI. Study protocol of a proposed Neurofeedback-Assisted Mindfulness Training Program on symptoms of anxiety and psychological distress associated with smartphone use in young adults: a randomized controlled trial. Front Public Health. 2024 Sep 4;12:1410932. doi: 10.3389/fpubh.2024.1410932. eCollection 2024. PMID 39296829